CLINICAL TRIAL: NCT03710343
Title: Metformin for Motor and Cognitive Improvement in Children With Cerebral Palsy: A Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MET-09-2017
Record Dates: First submitted 2018-07-11; First posted 2018-10-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Pediatric; Motor Function; GMFCS; Cognitive Function; Metformin
MeSH Terms: conditions — Cerebral Palsy | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The trial is designed as a 48 week limited institution two-site single case ABA study feasibility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Metformin oral tablet will be taken by mouth or through a gastrostomy tube, once or twice a day for 16 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Single case ABA study design. Phase B (intervention period) with metformin administered orally (or by gastrostomy tube) for 16 weeks.
  Other Names: Sandoz Metformin FC

SUMMARY:
The study design is a single-subject ABA clinical trial that is investigating the feasibility including adherence, safety and tolerability of metformin in children aged 5 to 18 years with cerebral palsy (CP). ABA refers to Phase A1 with no metformin, Phase B with metformin, and Phase A2 with no metformin. Secondarily, the study is exploring whether metformin has possible health benefits for improving motor function and cognition.

DETAILED DESCRIPTION:
The trial is designed as a 48 week limited institution two-site single case ABA study feasibility trial. ABA refers to Phase A1 with no metformin, Phase B with metformin, and Phase A2 with no metformin. Primary endpoints are feasibility, including recruitment, adherence to study medication and outcome measure completion, safety and tolerability of metformin. Key secondary endpoints are gross motor function and sustainability of intervention. Exploratory endpoints are cognitive and MRI measures as well as qualitative information regarding barriers to participation.

All participants will receive the study drug (metformin) during the 16 week intervention period.

This study will be done at two different locations in Toronto 1) Holland Bloorview Kids Rehabilitation Hospital and 2) the Hospital for Sick Children (SickKids). Each participant will be asked to go to both hospitals to do different tests and assessments for the study. Ten participants with physician diagnosis of CP age 5 to 18 with evidence of white matter imaging (WMI) or Grey Matter Imaging (GMI), and gross motor function classification system (GMFCS) levels II-V will be recruited for participation. MRI, cognitive testing and focus groups will be conducted at SickKids where paediatric protocols and processes have been developed.

ELIGIBILITY:
Inclusion criteria are as follows:

1. Physician diagnosis of cerebral palsy defined "as a group of permanent disorders of the development of movement and posture causing activity limitation that is attributed to non-progressive disturbances that occurred in the developing fetal or infant brain."
2. Evidence of WMI or GMI pattern on prior clinical neuro-imaging scanning (MRI)
3. No history of hypoglycemia after 2 years of age
4. No aspiration pneumonias in the last year requiring hospitalization
5. No lower extremity orthopedic surgery in the last six months prior to trial entry
6. No acute or chronic metabolic acidosis and/or lactic acidosis over the lifespan, including a lactate level greater than 2.4 mmol/L at the screening visit.
7. No history of renal disease
8. Age 5 to 18 years, 11 months at the time of enrollment
9. Either declare English as their native language or have had at least two years of schooling in English at the time of their baseline assessment
10. Gross Motor Function Classification System Level of II - V at the time of enrollment
11. Ability to communicate (verbal or non-verbal) pain or discomfort
12. With the exception of physiotherapy, no participation in active gross motor rehabilitation treatment (e.g. receiving lower extremity botulinum toxin injections, engaged in robotic walking therapy) up to 4 months prior to trial entry period and willingness to forgo introducing any new CP treatments during the 16 week trial period
13. Able to consume whole or crushed tablets swallowed orally or through a gastrostomy tube
14. Ability to understand and follow single step instructions/commands (i.e. blinking eyes, opening mouth, and moving head side to side).
15. Meet criteria for normal organ function requirements as described below:

Normal renal function defined as: Estimated glomerular filtration rate (eGFR) > 75ml/min/1.73m2

1. eGFR is calculated using the Schwartz formula: eGFR (mL/min/1.73 m²) = (0.41 × Height in cm) / Creatinine in mg/dL [29, 30]
2. Normal liver function defined as:

   * Total bilirubin < upper limit of normal (ULN) for age
   * SGOT (AST) or SGPT (ALT) < upper limit of normal (ULN) for age

Maximum AST Level (U/L) Male Female <12 years <47 <47

≥ 12 years <35 <30

Maximum ALT Level (U/L)

Male Female All Ages <50 <36

Maximum Total Billirubin Level ( μmol/L) Male Female

All Ages <20 <20

Informed consent (and assent, where applicable) will be obtained from the participants by study team members authorized to consent for this study

Exclusion criteria are as follows:

Participants who meet any of the following criteria will not be eligible to take part in the trial:

1. No prior clinically ordered neuro-imaging to allow determination of WMI or GMI
2. Have a known hypersensitivity to metformin hydrochloride or any of the excipients
3. Have Diabetes (Type I or II)
4. Have taken oral metformin previously
5. Have been part of another clinical intervention study within the past 3 months prior to study entry
6. Require sedation for blood tests
7. Treatment or planned treatment involving diuretics
8. Current or planned treatment with cationic drugs excreted by the kidneys (e.g. amiloride, cimetidine, digoxin, morphine, nifedipine, procainamide, quinidine, quinine, ranitidine, triamterene, trimethoprim and vancomycin).
9. Current or planned treatment with concomitant medications with potential unacceptable interaction with metformin including topiramate, lamotrigine, levetiracetam, beta blockers, ACE inhibitors, glycopyrrolate, and carbonic anhydrase inhibitors, or at the discretion of the delegated study physician for medications with potential interactions such as sertraline, lansoprazole and omeprazole.
10. Receiving deep brain stimulation or intrathecal baclofen
11. Dosage of oral baclofen and benzodiazepines stabilized for less than 2 months prior to study entry, and/or planning to change the dosage over the treatment period (if applicable)
12. Females who are pregnant, nursing, or planning a pregnancy during the study
13. Pernicious anemia (according to results of the screening visit blood draw)
14. Weight for age percentile less than 5%
15. Uncontrolled seizures with or without medication (defined by a seizure lasting longer than 10 minutes in duration within six months prior to study entry or change in seizure medication due to poor seizure control in the 3 months prior to trial entry).
16. History of congestive heart failure (including the use of diuretics) requiring pharmacologic treatment within two years prior to study entry

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
The first indicator of feasibility will be assessed | 1.25 years
  Whether 50% of identified eligible potential participants are consented.
The second indicator of feasibility will be assessed | 1.25 years
  Whether 80% of the study medication (metformin) was taken by all enrolled participants
The third indicator of feasibility will be assessed | 1.25 years
  Whether the GMFM-66 was performed for 80% of participants at all time points: pre-pre intervention , pre-intervention, post-intervention and at follow up (4 months post-intervention).
The fourth indicator of feasibility will be assessed | 1.25 years
  Whether an MRI was performed for 70% of participants at pre-intervention (i.e. beginning of the 16 week-intervention) and post-intervention (i.e. at the end of the 16-week intervention).
Tolerability and safety | 1.25 years
  Tolerability and safety of metformin will be evaluated with adverse event reporting and by semi-structured interviews of participants' perceptions of the study procedures known as the Safety Monitoring Uniform Research Form (SMURF) during the 16-week intervention period at all 7 safety visits.

SECONDARY OUTCOMES:
Gross Motor Function Measure-66 | Change in Gross Motor Function Measure-66 (GMFM-66) from pre-pre Intervention (visit 1) to baseline/pre-Intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  Gross motor function as assessed by the Gross Motor Function Measure-66 (GMFM-66).
Change in spasticity as measured by the Modified Tardieu Scale from baseline/pre-intervention (visit 2) to 48 weeks | Change in Modified Tardieu Scale (MTS) measure from baseline/pre-intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  Measured by the Modified Tardieu Scale (MTS), which consists of performing a passive muscle stretch at two velocities, slow and fast. The rater measures the angle of the spastic catch in the fast stretch (defined as R1) and then measures the passive range of motion during the slow stretch (defined as R2) in the ankle plantar flexors and knee flexors bilaterally. The difference between R2 and R1 will be the measure of the dynamic component of spasticity. Results are presented on a scale ranging from 0-4 where decreased scores indicate less resistance, which is considered to be a better outcome.

OTHER OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Change in CANTAB measures at different from from baseline/pre-intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  The CANTAB is a computerized test battery capable of capturing multiple data sources. Includes several tasks. Rapid Visual Information Processing: detection of target sequences of digits. Shorter reaction times indicate better information processing. Match to Sample Visual Search: matching test where the participant is shown a complex visual pattern and the participant must identify the matching box. More correct matching and shorter reaction times indicate better information processing. Simple Reaction Time: Measures simple reaction time. Shorter reaction times indicate better alertness and motor speed. Choice Reaction Time: Measures general alertness and motor speed. More correct responses and shorter reaction times indicate better alertness and motor speed.
NIH Toolbox (National Institutes of Health) | Change in NIH toolbox measures from from baseline/pre-intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  A computerized battery of tests that assesses cognitive function with standardized scores ranging from ages 3-85. Selected tests will assess executive function, processing speed, episodic memory, and working memory. Higher proportion of correct responses and reduced response times indicate better executive functioning, processing speed, episodic and working memory.
Children's Auditory Verbal Learning Test-2 [CAVLT-2] or Rey Auditory Verbal Learning Test [RAVLT] (depending on age of participant) | Change in CAVLT-2 measures from from baseline/pre-intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  The Children's Auditory Verbal Learning Test-2 [CAVLT-2] provides measures of immediate memory span as well as immediate and delayed recall. This will allow assessment of the extent of deficits within the areas of auditory verbal learning and memory. CAVLT-2 is applicable for children aged 6.6 to 17.11 years of age. As such, for this study, children between 5.0 to 6.5 years of age will not complete the CAVLT-2.
Wechsler Abbreviated Scale of Intelligence Second Edition [WASI-II] or Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition [WPPSI - IV], depending on the age of the participant. | Change in Wechsler Scales of Intelligence measures from baseline/pre-intervention (visit 2) to week 16 of Intervention (visit 9) to 48 weeks
  Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II) provides a brief measure of overall intelligence. WASI-II is applicable for people aged 6.0 to 90.11 years of age. For participants who are 5.0 to 5.9 years of age, the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI - IV) will be used instead
Changes in the tissue structure cortical-spinal tract and other relevant white matter tracts or grey matter tracts as measured by Diffusion Kurtosis Imaging (DKI). | Change in the tissue structure of cortical-spinal tract and other relevant white matter tracts or grey matter tracts from from baseline/pre-intervention (visit 2) to 32 weeks
  DKI is a magnetic resonance imaging (MRI) modality that measures water diffusion in the brain and provides information regarding tissue structure. Tractography will be used to identify the cortical-spinal tract and other relevant white matter tracts. Tractography defines white matter tracts based on regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Fehlings, MD, MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (2):
- Canada (2):
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No